CLINICAL TRIAL: NCT02259348
Title: CD45A-Depleted Haploidentical Hematopoietic Progenitor Cell and Natural Killer Cell Transplantation for Hematologic Malignancies Relapsed or Refractory Despite Prior Transplantation
Brief Title: Repeat Transplantation for Relapsed or Refractory Hematologic Malignancies Following Prior Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator's decision.
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REFNK1; NCI-2014-01925 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2016-09

CONDITIONS: Acute Lymphoblastic Leukemia (ALL); Acute Myeloid Leukemia (AML); Myeloid Sarcoma; Chronic Myelogenous Leukemia (CML); Juvenile Myelomonocytic Leukemia (JMML); Myelodysplastic Syndrome (MDS); Non-Hodgkin Lymphoma (NHL)
Keywords: Hematological malignancies; Allogeneic hematopoietic cell transplant; Refractory hematologic malignancy; Relapsed hematologic malignancy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Sarcoma, Myeloid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Juvenile; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Hematologic Neoplasms | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Granulocyte Colony-Stimulating Factor; Filgrastim; Interleukin-2; aldesleukin; Melphalan; Thiotepa; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participants (Experimental): Participants undergo a conditioning regimen with cyclophosphamide, fludarabine, aldesleukin (interleukin-2), natural killer cell therapy, anti-thymocyte globulin, rituximab, thiotepa, and melphalan prior to transplantation of T-cell depleted HPC transplant on day 0 and CD45RA-depleted HPC transplant on day 1. Beginning Day 6 post-transplant, patients receive G-CSF daily until ANC recovers to normal level.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: G-CSF; Biological: Interleukin-2; Drug: Melphalan; Drug: Thiotepa; Drug: Rituximab; Biological: Natural killer cell therapy; Biological: T-cell depleted HPC transplant; Biological: CD45RA-depleted HPC transplant

INTERVENTIONS:
Drug: Cyclophosphamide — Given intravenously (IV)
  Other Names: Cytoxan
Drug: Fludarabine — Given IV
  Other Names: Fludara; Fludarabine monophosphate
Biological: G-CSF — Given IV or subcutaneously (SQ)
  Other Names: Filgrastim; Neupogen®
Biological: Interleukin-2 — Given SQ
  Other Names: IL-2; Aldesleukin
Drug: Melphalan — Given IV
  Other Names: L-phenylalanine mustard; Phenylalanine mustard; L-PAM; L-sarcolysin; Alkeran®
Drug: Thiotepa — Given IV
  Other Names: ThioplexV; TESPA; TSPA
Drug: Rituximab — Given IV
  Other Names: Rituxan™
Biological: Natural killer cell therapy — Given IV
  Other Names: NK cell therapy
Biological: T-cell depleted HPC transplant — T-cell depleted hematopoietic stem cells will be infused on day 0.
  Other Names: HPC,A Infusion(ɑ/β T cell depleted)
Biological: CD45RA-depleted HPC transplant — CD45RA depleted stem cells will be infused on day 1.

SUMMARY:
This pilot phase II trial studies how well a new reduced intensity conditioning regimen that includes haploidentical donor NK cells followed by the infusion of selectively T-cell depleted progenitor cell grafts work in treating younger patients with hematologic malignancies that have returned after or did not respond to treatment with a prior transplant. Giving chemotherapy and natural killer cells before a donor progenitor cell transplant may help stop the growth of cells in the bone marrow, including normal blood-forming cells (progenitor cells) and cancer cells. It may also stop the patient's immune system from rejecting the donor's cells. When the healthy progenitor cells from a related donor are infused into the patient they make red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells (called graft-versus-host disease). Removing specific T cells from the donor cells before the transplant may prevent this.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

* To estimate engraftment by day +42 post-transplant in patients who receive CD45RA-depleted haploidentical donor progenitor cell transplantation following reduced intensity conditioning regimen that includes haploidentical natural killer (NK) cells.

SECONDARY OBJECTIVES:

* Estimate the incidence of malignant relapse, event-free survival, and overall survival at one-year post-transplantation.
* Estimate incidence and severity of acute and chronic (GvHD).
* Estimate the rate of transplant related mortality (TRM) in the first 100 days after transplantation.

Blood progenitor cells will be collected from adult donors to be used for transplantation. Donor cells will be processed and filtered in a laboratory at St. Jude using a machine called the CliniMACS™ device, and later infused (transplanted) into the participant through his/her veins.

Participants undergo a conditioning regimen beginning Day 21 prior to progenitor cell transplantation that includes chemotherapy medications and natural killer cells in preparation for transplantation. They will then receive T-cell depleted HPC transplant followed by CD45RA-depleted HPC transplant the following day.

ELIGIBILITY:
Inclusion Criteria:

* Age less than or equal to 21 years.
* One of the following hematologic malignancies that has relapsed or remains refractory after prior allogeneic hematopoietic cell transplant (HCT):

  * ALL, AML, Myeloid Sarcoma, CML, Juvenile myelomonocytic leukemia (JMML), myelodysplastic syndrome (MDS), non-Hodgkin lymphoma (NHL)
* Has a suitable single haplotype matched (≥ 3 of 6) family member donor.
* Does not have any other active malignancy other than the one for which this transplant is indicated.
* If prior central nervous system (CNS) leukemia, it must be treated and in CNS complete remission (CR)
* Does not have current uncontrolled bacterial, fungal, or viral infection.
* Patient must fulfill pre-transplant evaluation:
* Left ventricular ejection fraction > 40%, or shortening fraction ≥ 25%.
* Creatinine clearance (CrCl) or glomerular filtration rate (GFR) ≥ 50 ml/min/1.73m2.
* Forced vital capacity (FVC) ≥ 40% of predicted value; or pulse oximetry ≥ 92% on room air if patient is unable to perform pulmonary function testing.
* Karnofsky or Lansky (age-dependent) performance score ≥ 50 (See Appendix A).
* Bilirubin ≤ 3 times the upper limit of normal for age.
* Alanine aminotransferase (ALT) ≤ 5 times the upper limit of normal for age.
* Not pregnant. If female with child bearing potential, must be confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment.
* Not breast feeding
* DONOR: At least single haplotype matched (≥ 3 of 6) family member
* DONOR: At least 18 years of age.
* DONOR: HIV negative.
* DONOR: Not pregnant as confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment (if female).
* DONOR: Not breast feeding.
* DONOR: Regarding donation eligibility, is identified as either:

  * Completed the process of donor eligibility determination as outlined in 21 CFR 1271 and agency guidance; OR
  * Does not meet 21 CFR 1271 eligibility requirements, but has a declaration of urgent medical need completed by the principal investigator or physician sub-investigator per 21 CFR 1271.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Triplett, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve participants meeting eligibility criteria were enrolled at St. Jude Children's Research Hospital between November 2014 and February 2015.
Pre-assignment Details: Six enrolled participants were blood donors and did not undergo transplantation.
Period: Overall Study
Arm/Group | Participants
Started | 12
One Year Post-transplant | 2
Completed | 2
Not Completed | 10
Not completed — Donors | 6
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Arm/Group | Participants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.6 (5.5)
Age, Customized [Median (Full Range); unit: years]
  Age, Median | 12.2 [6.7 to 19.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Not otherwise specified Spanish, Hispanic, Latino | 1
  Non Spanish speaking, Non Hispanic | 5
Primary Diagnosis [Number; unit: participants] — AML = acute myeloid leukemia; MLL = myeloid-lymphoid leukemia; MDS = myelodysplastic syndrome
  participants
    AML with 11q23/MLL abnormalities | 2
    AML, multilineage dysplasia with prior MDS | 1
    AML, not otherwise specified | 2
    AML, without maturation | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Engrafted by Day 42 Post-transplant
Description: To estimate engraftment by day +42 post-transplant in patients who receive CD45RA-depleted haploidentical donor progenitor cell transplantation following reduced intensity conditioning regimen that includes haploidentical NK cells. Engraftment is defined as the first of 3 consecutive tests performed on different days of an ANC ≥ 500/mm^3 with evidence of donor cell engraftment.
Time Frame: Day 42 post transplantation
Measure: Number; unit: percentage of participants
Arm/Group | Participants
Number analyzed (Participants) | 6
percentage of participants | 100

2. Secondary Outcome: Incidence of Malignant Relapse
Description: The estimate of cumulative incidence of relapse will be estimated using Kalbfleisch-Prentice method. Death is the competing risk event. The number of participants with incidence of malignant relapse is given. Relapse was evaluated using standard WHO criteria for each disease.
Time Frame: one year post transplantation
Measure: Number; unit: participants
Arm/Group | Participants
Number analyzed (Participants) | 6
participants | 2

3. Secondary Outcome: Event-free Survival (EFS)
Description: The Kaplan-Meier estimate of event-free survival (EFS) along with their standard errors will be calculated using the SAS macro (bmacro251-Excel2007\kme) available in the Department of Biostatistics at St. Jude, where EFS = min (date of last follow-up, date of relapse, date of graft failure, date of death due to any cause) - date of transplant, and all participants surviving at the time of analysis without events will be censored. The number of participants who did not experience any of these events through one year post-transplant is given.
Time Frame: one year post transplantation
Measure: Number; unit: participants
Arm/Group | Participants
Number analyzed (Participants) | 6
participants | 2

4. Secondary Outcome: Overall Survival (OS)
Description: The Kaplan-Meier estimate of OS along with their standard errors will be calculated using the SAS macro (bmacro251-Excel2007\kme) available in the Department of Biostatistics at St. Jude, where OS = min (date of last follow-up, date of death) - date of transplant and all participants surviving at the time of analysis without events will be censored. The number of participants surviving to one-year post-transplantation is given.
Time Frame: one year post transplantation
Measure: Number; unit: participants
Arm/Group | Participants
Number analyzed (Participants) | 6
participants | 2

5. Secondary Outcome: Incidence and Severity of Acute GvHD
Description: The cumulative incidence of acute GvHD will be estimated using Kalbfleisch-Prentice method. Death is the competing risk event. The severity of acute GvHD. The number of participants with incidence by grade is given. Participants are graded on a scale from 1 to 4, with 1 being mild and 4 being severe.
Time Frame: 100 days post transplantation
Population: Two of six participants did not experience any acute GvHD.
Measure: Number; unit: participants
Arm/Group | Participants
Number analyzed (Participants) | 6
participants
  Grade I | 0
  Grade II | 0
  Grade III | 3
  Grade IV | 1

6. Secondary Outcome: Incidence and Severity of Chronic GvHD
Description: The cumulative incidence of chronic GvHD will be estimated using Kalbfleisch-Prentice method. Death is the competing risk event. The severity of chronic GvHD will be described. Chronic GvHD was evaluated using NIH Consensus Global Severity Scoring." The number of participants with incidence by severity is given.
Time Frame: one year post transplantation
Measure: Number; unit: participants
Arm/Group | Participants
Number analyzed (Participants) | 6
participants
  Mild | 0
  Moderate | 0
  Severe | 0

7. Secondary Outcome: Rate of Transplant-related Mortality (TRM)
Description: The cumulative incidence of transplant related mortality will be estimated using Kalbfleisch-Prentice method. Deaths before day 100 because of other reasons are the competing risk events.
Time Frame: 100 days post transplantation
Population: All six participants who received the protocol-defined treatment were evaluable for this analysis. One participant died of a non-transplant related cause (leukemia) prior to day 100. Although this participant did not complete the study to Day 100 post-transplantation, they were still evaluable for TRM.
Measure: Number; unit: participants
Arm/Group | Participants
Number analyzed (Participants) | 6
participants | 0

8. Post Hoc Outcome: Mean of Days to Absolute Neutrophil Count (ANC) Engraftment
Description: ANC engraftment is defined as the first of 3 consecutive tests performed on different days of an ANC ≥ 500/mm^3 with evidence of donor cell engraftment.
Time Frame: Day 42 post transplantation
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Participants
Number analyzed (Participants) | 6
days | 10.3 (1.03)

9. Post Hoc Outcome: Median Days to Absolute Neutrophil Count (ANC) Engraftment
Description: as for outcome 8
Time Frame: Day 42 post transplantation
Measure: Median (Full Range); unit: days
Arm/Group | Participants
Number analyzed (Participants) | 6
days | 10 [9 to 12]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from study enrollment through off-study date (up to 16 months).
Arm/Group | Participants
Serious Adverse Events (participants affected / at risk) | 5/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants (N=6)
Hemorrhage, pulmonary (Blood and lymphatic system disorders) | 1 (1)
Hepatic failure (disorder) (Hepatobiliary disorders) | 1 (1)
Infection, candida glabrata, GI tract (Infections and infestations) | 1 (1)
Infection, culture negative, sepsis (Infections and infestations) | 1 (1)
Infection, enterococcus faecalis, blood (Infections and infestations) | 1 (1)
Infection, escherichia coli, blood (Infections and infestations) | 1 (1)
Infection, klebsiella oxytoca, blood (Infections and infestations) | 1 (1)
Infection, pseudomonas aeruginosa, blood (Infections and infestations) | 1 (1)
Infection, staphylococcus epidermidis, blood (Infections and infestations) | 1 (1)
Infection, toxoplasmosis, cerebrospinal fluid (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Seizure (Nervous system disorders) | 2 (2)
Cryptogenic organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Failure, pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (disorder) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Failure, renal (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants (N=6)
Hypertension (Cardiac disorders) | 2 (4)
Hypotension (Cardiac disorders) | 3 (7)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 4 (4)
Pneumatosis (Gastrointestinal disorders) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 2 (2)
Hemorrhage, gastrointestinal (Gastrointestinal disorders) | 1 (1)
Abscess, mouth (Infections and infestations) | 1 (1)
Febrile neutropenia (Infections and infestations) | 5 (10)
Infection, adenovirus, respiratory tract (Infections and infestations) | 2 (2)
Infection, adenovirus, stool (Infections and infestations) | 3 (7)
Infection, BK virus, blood (Infections and infestations) | 1 (1)
Infection, BK virus, urine (Infections and infestations) | 1 (1)
Infection, candida albicans, oral mucosa (Infections and infestations) | 1 (1)
Infection, candida albicans, tracheostomy site (Infections and infestations) | 1 (1)
Infection, candida guilliermondii, blood (Infections and infestations) | 1 (1)
Infection, candida lusitaniae, small intestine (Infections and infestations) | 1 (1)
Infection, clostridium difficile, stool (Infections and infestations) | 1 (1)
Infection, coagulase negative staphylococcus, pleural fluid (Infections and infestations) | 1 (1)
Infection, disseminated fungus, organism unknown (Infections and infestations) | 1 (1)
Infection, enterobacter cloacae, trachael aspirate (Infections and infestations) | 1 (1)
Infection, human herpes virus 6, blood (Infections and infestations) | 3 (3)
Infection, rotavirus, stool (Infections and infestations) | 3 (3)
Infection, staphylococcus epidermidis, blood (Infections and infestations) | 1 (1)
Infection, upper respiratory (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Hallucinations (finding) (Nervous system disorders) | 1 (1)
Involuntary movement (finding) (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Bronchiolitis obliterans organizing pneumonia (disorder) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Infiltrates, pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Failure, renal (Renal and urinary disorders) | 1 (1)
Acute infusion reaction, boost (General disorders) | 1 (1)
Acute infusion reaction, granulocyte (General disorders) | 1 (1)
Acute infusion reaciton, NK cells (General disorders) | 1 (1)
Acute infusion reaction, stem cells (General disorders) | 1 (1)
Cytokine release syndrome, ATG (General disorders) | 3 (3)
Engraftment syndrome (General disorders) | 2 (2)
Systemic inflammatory response syndrome (disorder) (General disorders) | 1 (1)
Tumor lysis syndrome (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was terminated early due to investigator's decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes